CLINICAL TRIAL: NCT04779489
Title: Checkpoint Inhibitor and Radiation Therapy in Bulky, Node-Positive Bladder Cancer (CIRTiN-BC): A Phase II, Single-Arm Trial
Brief Title: Checkpoint Inhibitor and Radiation Therapy in Bulky, Node-Positive Bladder Cancer
Acronym: CIRTiN-BC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was closed to low accrual.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Solomon Woldu, Assistant Professor, Urology, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU-2021-0114
Record Dates: First submitted 2021-02-26; First posted 2021-03-03 (Actual); Results first posted 2023-08-22 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Bladder Cancer
Keywords: bladder cancer; lymph node metastasis; immunotherapy; radiation therapy
MeSH Terms: conditions — Urinary Bladder Neoplasms; Lymphatic Metastasis | interventions — DEAE-Dextran

STUDY DESIGN:
Intervention Model Description: single-arm interventional study
Masking Description: open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- PULSAR (Experimental): Eligible patients will receive next-generation stereotactic radiotherapy (PULSAR) 30-36 Gy in 3 fractions to the bladder and targetable, pathologically enlarged lymph nodes
  Interventions: Radiation: personalized ultrafractionated stereotactic ablative radiotherapy

INTERVENTIONS:
Radiation: personalized ultrafractionated stereotactic ablative radiotherapy — next-generation stereotactic ablative radiotherapy to bladder and enlarged lymph nodes
  Other Names: PULSAR

SUMMARY:
Clinically node positive (cN+) bladder cancer carries a poor prognosis, especially in patients who are unable to receive or fail to respond to neoadjuvant chemotherapy. Immune checkpoint inhibitor (ICI) therapy is FDA-approved in advanced bladder cancer for patients unable to receive or failing to respond to platinum-based chemotherapy. The present study seeks to determine if next-generation radiation therapy (personalized ultrafractionated stereotactic ablative radiotherapy, or PULSAR) is feasible and effective in patients receiving ICI for bulky cN+ bladder cancer.

DETAILED DESCRIPTION:
Patients are eligible for the trial if they have bulky, clinically node-positive (cN+) bladder cancer and have either recently initiated (within ≤ 1 week) or are planned to initiate immune checkpoint inhibitor (ICI) therapy due to either 1) ineligibility for/refusal of platinum-based downstaging chemotherapy; or 2) failure to achieve a complete clinical response to platinum-based downstaging chemotherapy. Patients will initiate PULSAR treatment 1-2 weeks after initiating ICI. PULSAR will be administered in 3 fractions of 12 Gy each (36 Gy total) at 12-16 day intervals and patients will undergo radical cystectomy with bilateral extended pelvic lymph node dissection within 4-8 weeks after completion of PULSAR. ICI therapy will be administered according to the FDA-approved dosing route and schedule and will be continued during PULSAR treatments.

PULSAR treatment will be initiated 1-2 weeks after the patient is initiated on an FDA-approved ICI agent. PULSAR will be administered in 3 fractions of 12 Gy each at 12-16 day intervals. Target areas will include the region of the bladder containing the primary tumor (confirmed, if necessary, on office flexible cystoscopy at UTSW) and to up to five targetable, pathologically enlarged bulky lymph nodes (as deemed feasible by the treating radiation oncologist). Non-enlarged pelvic lymph nodes will be spared to minimize adverse effects on the tumor immune response.

ELIGIBILITY:
Inclusion Criteria

* Bladder cancer, confirmed pathologically on transurethral resection of bladder tumor (TURBT) or on bladder biopsy. Pure urothelial, variant urothelial, or any proportion of squamous cell carcinoma are permitted. Questions about eligibility may be resolved by consultation with UTSW pathology but formal pathologic review is not required.
* Bulky, clinically node positive disease (cN+) defined as: 1) a single pelvic lymph node of ≥ 1.5 cm largest diameter on CT or MRI; or 2) multiple pelvic lymph nodes ≥ 1 cm largest diameter on CT or MRI. Pathologic confirmation is not required. Imaging to establish eligibility must have been obtained no more than 60 days prior to trial enrollment. The scans must be personally reviewed by the enrolling clinician. For imaging studies obtained outside of UT Southwestern, imaging review of node status and sign off by the enrolling investigator is required. Review and sign off by a UTSW radiologist is optional in ambiguous or questionable cases, but is not mandatory.
* Age ≥ 18 years.
* ECOG performance status 0-1.
* Appropriate candidate for radical cystectomy, as determined by the treating urologist.
* Appropriate candidate for stereotactic ablative radiotherapy, as determined by the treating radiation oncologist.
* Patient is planned to initiate or is within 1-3 weeks of initiation of FDA-approved immune checkpoint inhibitor therapy based on ineligibility to receive platinum-based downstaging chemotherapy (DCT) (Cohort 1, as detailed below) or failure to achieve clinical complete response to platinum-based DCT (Cohort 2, as detailed below).

Cohort 1 (chemotherapy-ineligible) - either of:

* patient staged with bulky cN+ disease as defined above, medically ineligible to receive any platinum-based chemotherapy or, after appropriate and documented counseling, refusing to receive any-platinum-based chemotherapy; or
* patient staged with bulky cN+ disease as defined above, medically ineligible to receive cisplatin-based chemotherapy, with PD-L1 positive tumor (according to methodology described in the FDA approval label for the respective ICI agent)

Cohort 2 (chemotherapy non-responding) - any of:

* patient, initially staged with bulky cN+ disease as defined above, with radiologic progression after two cycles of platinum-based DCT (per RECIST 1.1 criteria: ≥20% increase in summed short-axis diameter of visible lesions with ≥ 5 mm absolute increase)
* patient, initially staged with bulky cN+ disease as defined above, failing to achieve radiologic complete response after three or four cycles of platinum-based DCT (failure of all enlarged lymph nodes to decrease to < 1 cm short-axis diameter)
* patient, initially staged with bulky cN+ disease as defined above, failing to achieve radiologic complete response after one or two cycles of platinum-based DCT which was discontinued due to patient intolerance
* patient, initially not staged with bulky cN+ disease as defined above, who progresses to cN+ disease as defined above after two or more of cycles of platinum-based DCT
* Permitted downstaging chemotherapy regimens are gemcitabine/cisplatin (gem/cis), gemcitabine/carboplatin (gem/carbo), and methotrexate/vinblastine/doxorubin/cisplatin (MVAC, in any dose variant).
* Permitted immune checkpoint inhibitor agents are those FDA-approved for platinum-ineligible (Cohort 1) or platinum-refractory (Cohort 2) bladder cancer: atezolizumab or pembrolizumab for Cohort 1; atezolizumab, avelumab, nivolumab, or pembrolizumab for Cohort 2. If additional immune checkpoint inhibitor (anti-PD1, anti-PD-L1, and/or anti-CTLA4) agents are approved for use in advanced urothelial carcinoma during the study, these agents will be permitted as well.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria

* Medical or anatomic contraindication to any of the study treatment modalities (radical cystectomy, stereotactic ablative radiotherapy, immune checkpoint inhibitor therapy).
* Non-urothelial histology (other than pure squamous cell, which is permitted) including pure adenocarcinoma, pure small cell carcinoma, sarcoma, lymphoma, non-genitourinary primary (e.g. colorectal).
* Metastatic (cM1) disease, defined as 1) lymph nodes ≥ 1 cm above the aortic bifurcation (cM1a), or metastases to bone, brain, or any visceral site (cM1b). Patients with a single enlarged retroperitoneal lymph node will be eligible with an adequately performed lymph node biopsy showing no metastatic disease or with a PET scan showing absence of FDG avidity.
* Second primary malignancy, except: 1) non-metastatic (cM0) prostate cancer, 2) non-metastatic (cM0) endometrial cancer, 3) non-melanoma skin cancer, 4) cervical squamous cell carcinoma in situ, 4) any AJCC Stage I/II or organ-confined primary malignancy for which the patient has undergone curative treatment and has been without evidence of disease for three years.
* Prior pelvic radiation therapy.
* Autoimmune disease rendering the patient ineligible for ICI.
* Treatment with any immunosuppressive agent within 14 days of study entry, excluding topical or inhaled corticosteroids or adrenal-replacement steroids.
* End stage renal disease requiring dialysis.
* HIV infection, unless stable on HAART with CD4+ count > 400.
* Subjects may not be receiving any other investigational agents for the treatment of the cancer under study.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to atezolizumab, avelumab, durvalumab, nivolumab, pembrolizumab, or other agents used in study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia (other than atrial fibrillation / atrial flutter), or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirements.
* Subjects must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2023-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Solomon L Woldu, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PULSAR
Started | 1
Completed | 0
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | PULSAR
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Protocol Completion
Description: proportion of patients completing PULSAR and undergoing radical cystectomy
Time Frame: 16 weeks
Population: One subject was enrolled and completed therapy but before the last two visits were completed, the study was terminated. Not enough data was collected to be analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | PULSAR
Number analyzed (Participants) | 1
Participants | 1

2. Secondary Outcome: Progression-free Survival
Description: proportion of patients without disease progression
Time Frame: 2 years
Population: One subject was enrolled and completed therapy. They study was terminated before the last two visits were completed and data could not be collected to be analyzed.
Arm/Group | PULSAR
Number analyzed (Participants) | 0

3. Other Pre Specified Outcome: Major Complication Rate
Description: patients experiencing Clavien-Dindo Grade III+ surgical complication
Time Frame: 90 days
Population: One subject was enrolled and completed therapy. They study was terminated before the last two visits were completed. Not enough data was collected to be analyzed.
Arm/Group | PULSAR
Number analyzed (Participants) | 0

4. Other Pre Specified Outcome: Pathologic Complete Response
Description: patients achieving pathologic ypT0 N0 status
Time Frame: at time of radical cystectomy
Population: as for outcome 3
Arm/Group | PULSAR
Number analyzed (Participants) | 0

5. Other Pre Specified Outcome: Pathologic Non-muscle Invasive Downstaging
Description: patients achieving pathologic ≤ ypT1 N0 status
Time Frame: at time of radical cystectomy
Population: as for outcome 3
Arm/Group | PULSAR
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Pathologic Organ-confined Downstaging
Description: patients achieving pathologic ≤ ypT2 N0 status
Time Frame: at time of radical cystectomy
Population: as for outcome 3
Arm/Group | PULSAR
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Pathologic Complete Nodal Response
Description: patients achieving pathologic ypN0 status
Time Frame: at time of radical cystectomy
Population: as for outcome 3
Arm/Group | PULSAR
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Residual Disease at Surgery
Description: patients with microscopic (R1) or gross (R2) residual disease
Time Frame: at time of radical cystectomy
Population: as for outcome 3
Arm/Group | PULSAR
Number analyzed (Participants) | 0

9. Other Pre Specified Outcome: Ureteroenteric Stricture Rate
Description: proportion of patients requiring procedural intervention for ureteroenteric stricture
Time Frame: 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year, 5 months
Arm/Group | PULSAR
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PULSAR (N=1)
Fever (General disorders) | 1 (2)
Pyelonephritis (Renal and urinary disorders) | 1 (1)
Worsening Falling /Unsteadiness (Nervous system disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (2)
Intra-Abdominal Abscess (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PULSAR (N=1)
Dry Mouth (Gastrointestinal disorders) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Adrenocorticotropic Hormone Level <5 (Endocrine disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Elevated Liver Function Test (Infections and infestations) | 1 (1)
Draining from abdomen (Gastrointestinal disorders) | 1 (2)
Pain to testicles (Reproductive system and breast disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-09): https://cdn.clinicaltrials.gov/large-docs/89/NCT04779489/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/89/NCT04779489/ICF_001.pdf